CLINICAL TRIAL: NCT01612754
Title: Noise Reduction Programme by Work Rules and Technical Devices (i.e.SoundEar-TM)for Surgical Theathres
Brief Title: Prospective Trial on Noise Reduction in Surgical Operating Theaters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: University of Zurich (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Carsten Engelmann, Oberarzt Kinderchirurgie, Hannover Medical School
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: SA 02
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Efficacy of a Noise Reduction Program; Surgical Complications; Sound Pressures in the Operating Theatre
Keywords: Reduction of noise pollution; Specifically enforced workplace rules; Stress; Sound Ears (TM); Error

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reference group - cloaked noise meters (No Intervention): Reference group or phase 1
  Theatre equipped with multiple sound meters disguised as CO2 meter for sound probing in the absence of a research clerk with personnel completely unaware of sound measurements.
- Control Noise AND Stress measurements (Sham Comparator): Control Group - Phase 2
  No intervention but research clerk is present in theatre to protocoll the operation and test for stress by collecting saliva cortisol and probing electrodermal activity
  Interventions: Behavioral: Presence of an examiner in the concerned theatre
- Noise Reduction Intervention Group (Experimental): Intervention Group - Phase 3
  A panel of noise reduction measures (staff workplace rules, technical devices as optical noise warners, optical telephones) is put into effect. Surgeons are monitored by biometry, psychometry and the outcome.
  Interventions: Behavioral: Noise reduction work place rules

INTERVENTIONS:
Behavioral: Noise reduction work place rules — Information conferences for all theatre staff (100%)on the detrimal effects of high noise levels in the operating theatre. Issue of "workplace rules" on handouts and poster on theatre doors: Ban of all mobile phones from theatre. Only conversations about the ongoing case are allowed. No restocking etc. during an operation and no work in this operating room concerning other patients (e.g. later on the list). Turnig of of unnecessary suckers, warming devices etc. . No in and out during the procedure.
  Technical: Sound Ears (TM, Sound Ear A.S. Copenhagen, Denmark) taped to all 4 Walls. Optical Telephones.
  Other Names: Sound Ears (TM, Sound Ear A.S. Copenhagen, Denmark)
  Arms: Noise Reduction Intervention Group
Behavioral: Presence of an examiner in the concerned theatre — Research Clerk present in theatre, writes on note pad.
  Arms: Control Noise AND Stress measurements

SUMMARY:
Aim of Study: Adverse effects from noise pollution in operation theatres have been throughly demonstrated. We assessed the impact of a noise reduction program in paediatric surgery.

Methods: A prospective controlled study on 156 operations performed by 16 surgeons was conducted. The sound levels before and after a noise reduction program based on education, rules and technical devices (Sound Ear tm) were assessed. Endpoints were spatially resolved sound levels matched by the surgeon's biometric (saliva cortisol, electrodermal activity) and behavioural stress responses (questionnaires). These were correlated with mission protocols and NoiSeQ for individual noise sensitivity.

DETAILED DESCRIPTION:
We recorded median noise levels in the control vs. interventional group including the count of peak events with different tresholds.

Three phases were conducted: 1. Reference group/phase I 2. Control group/phase II The full data set was recorded by a research clerk present in theatre however all staff were left unaware of the study purpose 3. Intervention group/phase III. The intervention consisted of a panel of work rules including mainly communication regulations (only conversations concerning the current case were allowed, no in and out during surgery, mobile phone ban etc.. Measures were backed by intervention conferences, posters and pictograms. .

A wear off-effect was sought after . Biometrically, we analyzed the surgeon's pre- to postoperative rise in cortisol and the proportion of the surgeon's electrodermal potentials of >15µS indicating severe stress. Intra-team communication, a decrease in disturbing conversations and sudden noise peaks were investigated and correlated with the individual noise sensitivity determined by the noise Q questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* all operations of our tertiary referral center practice of the regular day programme involving children from preterm babies up to children of 16 years of age including emergencies at regular hours with a duration of > 20 mins and < 5 hours

Exclusion Criteria:

* After hour emergency surgery
* Pediatric surgery cardiac cases
* surgeries <20 mins/>5hrs

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Noise level (dB(A)) in the operation room at the surgeon's place | continous during operation
  noise levels are sampled simultaneously at 4 point (surgeon, nurses 1+2 and anestesiology workplace

SECONDARY OUTCOMES:
Surgeons intraoperative biometric and psychometric stress response | before, during and after operations
  Surgeons Cortisol Levels and Electrodermal activity are measured as he/she is submitted to questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten R Engelmann, MD, PhD, Principal Investigator — Hannover Medical School, Germany
Locations (1):
- Pediatric Surgery Department, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Conrad C, Konuk Y, Werner PD, Cao CG, Warshaw AL, Rattner DW, Stangenberg L, Ott HC, Jones DB, Miller DL, Gee DW. A quality improvement study on avoidable stressors and countermeasures affecting surgical motor performance and learning. Ann Surg. 2012 Jun;255(6):1190-4. doi: 10.1097/SLA.0b013e318250b332. PMID 22584632
- [Background] Engelmann C, Schneider M, Kirschbaum C, Grote G, Dingemann J, Schoof S, Ure BM. Effects of intraoperative breaks on mental and somatic operator fatigue: a randomized clinical trial. Surg Endosc. 2011 Apr;25(4):1245-50. doi: 10.1007/s00464-010-1350-1. Epub 2010 Sep 11. PMID 20835716
- [Background] Shapiro RA, Berland T. Noise in the operating room. N Engl J Med. 1972 Dec 14;287(24):1236-8. doi: 10.1056/NEJM197212142872407. No abstract available. PMID 5084988
- [Background] Moorthy K, Munz Y, Undre S, Darzi A. Objective evaluation of the effect of noise on the performance of a complex laparoscopic task. Surgery. 2004 Jul;136(1):25-30; discussion 31. doi: 10.1016/j.surg.2003.12.011. PMID 15232535
- [Background] Connor A, Ortiz E. Staff solutions for noise reduction in the workplace. Perm J. 2009 Fall;13(4):23-7. doi: 10.7812/TPP/09-057. PMID 20740099
- [Background] Arora S, Hull L, Sevdalis N, Tierney T, Nestel D, Woloshynowych M, Darzi A, Kneebone R. Factors compromising safety in surgery: stressful events in the operating room. Am J Surg. 2010 Jan;199(1):60-5. doi: 10.1016/j.amjsurg.2009.07.036. PMID 20103067